CLINICAL TRIAL: NCT06860880
Title: Combating Cancer-Related Fatigue: A Personalized Supportive Care Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: CLL Society (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2403
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Indolent Lymphomas; Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Lymphoplasmacytic Lymphoma; Waldenstrom Macroglobulinemia; Cutaneous T Cell Lymphoma
Keywords: exercise; dietary intervention
MeSH Terms: conditions — Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Cutaneous; Motor Activity | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who are with chronic lymphocytic leukemia/small lymphocytic lymphoma (Other): Patients who are with chronic lymphocytic leukemia/small lymphocytic lymphoma were assessed and received exercise and diet programs.
  Interventions: Other: Exercise; Other: Diet

INTERVENTIONS:
Other: Exercise — Each patient will receive an individualized exercise prescription that will encompass both aerobic and resistance training, with modifications as necessary to accommodate each patient's needs, abilities, and medical condition. For those not participating in any formal exercise at baseline, the exercise prescription will consist of a basic conditioning program targeting 150 minutes of moderate physical activity weekly with the assistance of a physical therapist if deemed appropriate.
Other: Diet — Participants will undergo nutritional consultations with a registered dietitian who specializes in oncology. The dietitian will provide tailored dietary recommendations using evidence-based nutrition guidelines. Participants will also be screened ffor ormal nutrition based on American Society for Parenteral and Enteral Nutrition (ASPEN) guidelines as indicated.

SUMMARY:
This health services study will assess a multidisciplinary intervention program directed at fatigue mitigation among patients diagnosed with indolent lymphomas. Specifically, 30 subjects with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) and 10 subjects with Follicular Lymphoma (FL), marginal zone lymphoma (MZL), lymphoplasmacytic lymphoma (LPL), Waldenström's Macroglobulinemia, or Cutaneous T Cell Lymphoma (CTCL) will be included.

DETAILED DESCRIPTION:
All subjects will be assigned to an exercise and dietary intervention program. Patients will engage in two patient-clinician consultations for exercise and nutrition. The individualized exercise plan designed based on the subject's medical history, current exercise habits, and specific needs, will include a mix of aerobic and resistance training.

Concurrently, participants will receive nutritional consultations from a specialized oncology dietitian. These sessions will focus on creating a diet plan tailored to each participant's nutritional needs, considering their treatment and overall health. Study participants will complete weekly exercise journals to track adherence to the exercise prescription and complete weekly assessments of their adherence to dietary recommendations on an integer scale ranging from 0-10.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

* Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
* Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* Confirmed diagnosis of indolent lymphoma, Waldenström's Macroglobulinemia, or Cutaneous T Cell Lymphoma.
* Significant symptoms of fatigue, as defined by PROMIS Fatigue score >50.

Exclusion Criteria:

* Other co-existing malignancies.
* Significant cognitive impairment as defined by Mini-Cog score 0-2 (out of 5) that would prevent understanding of assessments or interventions.
* Unstable or serious illness (e.g., unstable cardiac arrhythmia, severe anemia/thrombocytopenia) that would prevent safe participation in an exercise regimen, per the discretion of the treating physician.
* Individuals who are not able to consume an oral diet, due to swallowing difficulties or other reasons, as this might interfere with the nutritional intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of consented patients who are referred | Baseline
  The proportion of consented patients with chronic lymphocytic leukemia (CLL) or other forms of indolent lymphoma who are referred to cancer rehabilitation and dietician and attend an initial appointment with each.

SECONDARY OUTCOMES:
Overall acceptability | Baseline and post-3 months follow-up
  Overall acceptability will be measured as the proportion of participants who report being "Neutral," "Satisfied" or "Very Satisfied" with the intervention utilizing the Cancer Fatigue Program Participant Feedback Questionnaire- Part 1. The questionnaire has 2 parts and the first part has 8 multiple choice questions. Options are very Dissatisfied, Dissatisfied, Neutral, Satisfied, Very Satisfied.
Differences in self-reported fatigue | Baseline and post-3 months follow-up
  Differences in self-reported fatigue will be determined by the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue (PROMIS Item Bank v1.0 Fatigue Short Form13a (FACIT-Fatigue)) questionnaire. It uses a scoring system to assess the severity of fatigue and its impact on daily activities. There are 13 items and each item in the short form has five response options, typically ranging from 1 (not at all) to 5 (very much), the lowest possible raw score is 13, and the highest possible raw score is 65.
Differences in overall health | Baseline and post-3 months follow-up
  Differences in overall health will be determined by Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health (PROMIS Scale v1.2 Global Health) scores. The PROMIS Scale v1.2 Global Health measures both physical and mental health through a set of items. Each item has five response options, typically ranging from 1 (poor) to 5 (excellent). Higher Scores: Indicate better health and lower Scores: Indicate poorer health.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Jensen, MD MSCR, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Basnight Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials